CLINICAL TRIAL: NCT04689542
Title: Effects of Surgical Face Mask on Submaximal Exercise Test in Patients With COVID-19
Brief Title: Surgical Face Mask Effects in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Poncin, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: COSIT
Record Dates: First submitted 2020-12-29; First posted 2020-12-30 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: Sit-To-Stand test; Surgical Facemask; Dyspnea
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Facemask (Experimental): The surgical facemask will be worn during the sit-to-stand test
  Interventions: Other: Sit-To-Stand test
- Control (No Intervention): No facemask will be worn during the sit-to-stand test

INTERVENTIONS:
Other: Sit-To-Stand test — The 1-minute sit-to-stand test will be realized with or without a surgical facemask covering the face of the patient with COVID-19
  Arms: Surgical Facemask

SUMMARY:
The use of personal protective equipment is mandatory for healthcare workers caring patient with COVID-19. To maximise the reduction of virus spread during clinical procedures involving the presence of healthcare workers, it is also recommended to patients to wear surgical facemask. Routine clinical procedures include cardio-pulmonary and strengthening exercises. During these exercises, the wearing of a face mask may be difficult to tolerate by patients, especially since they experience breathing difficulties due to the illness. Therefore, this study aims to verify the effects of the surgical facemask on breathing difficulties and exercise performance during a 1-minute sit to stand test.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for COVID-19
* No need of supplemental oxygen during the procedure

Exclusion Criteria:

* Altered state of consciousness
* Respiratory co-morbidities
* Neurological or orthopedic co-morbidities susceptible to alter the reliability of the sit-to-stand test
* Having required high flow nasal cannula or non-invasive ventilation during the hospital stay

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Changes in dyspnea level | Before, immediately after and 2 minutes after the sit-to-stand test
  The Modified Borg dyspnea scale will be used to estimate dyspnea This scale range from 0 (no dyspnea) to 10 (maximal dyspnea)

SECONDARY OUTCOMES:
Changes in respiratory rate | Before, immediately after and 2 minutes after the sit-to-stand test
  Respiratory rate will be measured using two inductive plethysmography belts
Changes in heart rate | Before, immediately after and 2 minutes after the sit-to-stand test
  Heart rate will be measured using a pulse oximeter
Changes in pulsed oxygen saturation (SpO2) | Before, immediately after and 2 minutes after the sit-to-stand test
  SpO2 will be measured using a pulse oximeter
Number of sit-to-stand repetition | 1 minute
  The number of repetitions will be manually counted

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium